CLINICAL TRIAL: NCT03221894
Title: A Retrospective Study to Investigate the Additive Effectiveness of Chinese Herbal Medicine in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Beijing Hospital (Other Government); Chinese PLA General Hospital (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Prof., Dongzhimen Hospital, Beijing
Other Study IDs: 2017-IRT-0810
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
Keywords: Complementary therapies
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional therapy with herbs: Patients were treated with conventional therapy with Chinese herbal medicine (GRAPE granules).
  Interventions: Dietary Supplement: GRAPE granules
- Conventional therapy alone: In conventional therapy group, donepezil was the commonly used ChEI(cholinesterase inhibitor) to treat mild to severe AD patients. Memantine, a NMDA(N-methyl-D-aspartate ) antagonist, was given to moderate and severe AD patients. The dose of donepezil ranged from 5 to 10 mg once a day according to patients.

INTERVENTIONS:
Dietary Supplement: GRAPE granules — GRAPE granules was mainly consisted of herbal medicines: Ren Shen (Ginseng, 10g/d), Di Huang (Rehmannia glutinosa, 30g/d), Shi Cangpu (Acorus tatarinowii, 10g/d), Yuan Zhi (Polygala tenuifolia, 10g/d), Yin Yanghuo (Epimedium brevicornu, 10g/d), Shan Zhuyu (Cornus officinalis, 10g/d), Rou Congrong (Cistanche deserticola, 10g/d), Yu Jin (Curcuma aromatica, 10g/d), Dan Shen (Salvia miltiorrhiza, 10g/d), Tian Ma (Angelica sinensis, 10g/d), Tian ma (Gastrodia elata, 10g/d), and Huang Lian (Berberine, 10g/d), which were supplied by Beijing Tcmages Pharmaceutical Co., LTD, Each bag of granules with 150ml warm water melt was taken orally twice a day.
  Groups: Conventional therapy with herbs

SUMMARY:
In China, herbal therapy as a complementary therapy is very popular. Should conventional therapy (such as donepezil and memantine) combined with herbal therapy make add-on benefit? Cognition, activities of daily living and behavioral symptoms will be assessed. Data will be collected from the medical records of patients with Alzheimer's disease (AD) in memory clinics.

DETAILED DESCRIPTION:
Conventional therapy (CT), such as donepezil and memantine are well- known short-term treatments for the symptoms of Alzheimer's disease (AD). The efficacy of them, however, drops below baseline level after 9 months. Should Chinese herbal medicine make add-on benefit? The GRAPE formula was designed by Prof. J Tian, a prepared granules of Chinese herbs, according to Qifuyin in Jing Yue Quan Shu (published in A.D. 1624). Patients treated with CT+herbal therapy or CT alone for up to and over 12 months are collected. Cognition, activities of daily living and behavioral symptoms are selected as outcomes for assessing the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in cognitive functions for a period greater than 6 months;
* Objective evidence of significantly impaired episodic memory together with at least one of other cognitive domains on testing;
* Global cognitive decline measured by mini-mental state examination (MMSE) adjusted for education: ≤22 for illiteracy, ≤23 for primary school, ≤24 for middle school,≤26 for high education;
* Impaired abilities of daily living, ADLs score ≥16;
* Clinical Dementia Rating (CDR) total score 0.5~3.0;
* ≤4 point on Hachinski Ischaemic Score (HIS);
* Age-adjusted medial temporal lobe atrophy scale (MTA-scale) based on coronary magnetic resonance imaging (MRI) scan of the brain (1.0 or more for ≤65 years; 1.5 or more for ≤75 years and 2.0 or more for ≥75 years);
* Other causes of dementia excluded.

Exclusion Criteria:

* Sudden onset of cognitive disorder with focal nervous system signs in the early stages of disease, (e.g., incomplete paralysis, anesthesia, dysfunctional visual field, and dystaxia);
* Early occurrence of the following symptoms: gait disturbances, seizures, extrapyramidal signs, hallucinations and cognitive fluctuations;
* Any major psychiatric disorders (e.g., DSM-IV(Diagnostic and Statistical Manual of Mental Disorders) defined psychosis, major depression, bipolar disorder, or alcohol or substance abuse);
* Other conditions that may explain cognitive impairment (e.g., hypothyroidism, electrolyte imbalance, toxic, inflammatory, and metabolic disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD patients involved in this retrospective, observational study will be selected from the clinic registration system of memory clinics in Beijing. All the participants underwent routine clinical assessments, including detailed medical history, cognitive and neuropsychological tests, neurological examinations, laboratory tests (i.e. thyroid function, folic acid levels, vitamin B12 levels, and routine blood tests), and neuroimaging. Participants with detailed medical history will be sampled and grouped into two cohorts according the therapies received.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Up to 12 months, repeated measurement every 3 months.
  Change of global cognition was measured by MMSE, a 30-point scale, higher score indicates better cognition.

SECONDARY OUTCOMES:
Activities of Daily Living (ADLs) | Up to 12 months, repeated measurement every 3 months.
  Both basic ADLs (6-items) and instrumental ADLs (8-items) were measured. The ADLs contain 14 items (score 1-4), the range is 14 to 56, and higher scores indicate worse function.
Clinical Dementia Rating (CDR) | Up to 12 months, repeated measurement every 3 months.
  The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias. 0 = Normal, 0.5 = Very Mild Dementia, 1 = Mild Dementia, 2 = Moderate Dementia, 3 = Severe Dementia.
Neuropsychiatric Inventory (NPI) | Up to 12 months, repeated measurement every 3 months.
  NPI was used for rating the behavioral and psychological symptoms of dementia (BPSD), including 12-items, with a score rang from 0-144, higher score indicates worse state.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou TIAN, Dr, Principal Investigator — Dongzhimen Hospital, BUCM
Locations (1):
- Dongzhimen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets are available from the PI on reasonable request.